CLINICAL TRIAL: NCT05446948
Title: Comparison of the Efficacy of Standard 25 Gauge (25G)+ and Beveled 27 Gauge (27G)+ Vitrectomy Systems in Proliferative Diabetic Retinopathy
Brief Title: Observation of the Efficacy of Different Vitrectomy Systems to Treat Proliferative Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Principal Investigator, Zhenchuan Zheng, Principal investigator, Tianjin Medical University Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021KY-27
Record Dates: First submitted 2022-06-29; First posted 2022-07-07 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Proliferative Diabetic Retinopathy; Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- beveled 27G+ group (Experimental): The group of patients underwent vitrectomy with a beveled 27G+ vitrectomy system.
  Interventions: Device: beveled 27G+ vitrectomy system
- 25G+ group (Active Comparator): The group of patients underwent vitrectomy with a standard 25G+ vitrectomy system.
  Interventions: Device: standard 25G+ vitrectomy system

INTERVENTIONS:
Device: beveled 27G+ vitrectomy system — The device is a novel 27G+ vitrectomy system, whose probe tip is beveled.
  Arms: beveled 27G+ group
Device: standard 25G+ vitrectomy system — The device is a traditional instrument, and its probe tip is flat.
  Arms: 25G+ group

SUMMARY:
In recent years, vitrectomy has moved toward a minimally invasive vitrectomy surgery (MIV) system, which could effectively reduce the occurrence of operation complications, while reducing the time of post-operation recovery.

With an improved design of bevel tip and a high cutting rate capacity of 10000cpm, Advanced ULTRAVIT® probes potentially provide an strong technical support for the application of MIV. The new probe facilitates great control during delicate surgical maneuvers, such as separating the hyaloid from the retinal surface, dissecting fibrovascular tissue off the surface of retina.

However, there was no sufficient clinical evidence to support the benefits of Advanced ULTRAVIT ® probes in the complicated vitreoretinal surgery, such as proliferative diabetic retinopathy. More importantly, there is an urgent need of clinical evidence to support 10000cpm launch and conversion which is major objective of 2021 VR growth strategies.

DETAILED DESCRIPTION:
This exploratory study, aiming to demonstrate the beneficial of 27 Gauge probe, which can be flexibly applied as a multifunctional tool for membrane removal by reducing frequencies of switching device, reducing the traction to eyeball during device entering and leaving the eye. Moreover, the outcomes from this study would be an strong evidence to support further comparative study to comprehensively demonstrate the superior function compare to current heavily used 5K 25 gauge probe.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with vitreous hemorrhage and tractional retinal detachment (TRD) confirmed by fundus image and B ultrasound examination, consistent with the diagnosis of severe proliferated diabetic retinopathy (PDR).
2. Patient that could follow up postoperatively at the clinic for 6 months more.
3. All the surgeries were performed by one well-experienced retinal surgeon.

Exclusion Criteria:

1. Corneal lesions affecting operative field, such as corneal opacity or scar; History of vitreoretinal surgery;
2. External eye infections;
3. History of systemic thromboembolism;
4. Uncontrolled hypertension or hyperglycemia;
5. Coagulation abnormalities or currently using anticoagulant drugs other than aspirin;
6. Unable to meet postoperative position requirements;
7. Unable to be followed up regularly.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
the convenience in operating | during surgery
  The convenience will be indicated by times of ancillary instrument using, which evaluated based on the recorded surgical video.
the efficiency of stripping membrane | during surgery
  It will be measured by the area of membrane removed per minute by probe.

SECONDARY OUTCOMES:
best corrected visual acuity (BCVA) | baseline to 6 months post-surgery
  BCVA using a logMAR visual acuity chart method

OTHER OUTCOMES:
intra-surgery complications | during surgery
  The complications include hemorrhage, iatrogenic retinal breaks, iatrogenic cataracts and occurrence of hypotony during the surgery. They can be detected by a microscope during surgery.
Post-operative complications | within 6 months after surgery
  The complications include recurrent vitreous hemorrhage, retinal detachment, re-operation and ocular hypertension. They can be detected through ophthalmoscope, fundus image, B ultrasound, ophthalmotonometer and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Li, Principal Investigator — Tianjin Medical University Eye Hospital
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No